CLINICAL TRIAL: NCT00985270
Title: PXR-agonisti Rifampisiinin Vaikutukset Glukoosi-, Lipidi- ja Hormonihomeostaasiin
Brief Title: Pregnane X Receptor (PXR) Agonist Rifampicin Effects on Glucose, Lipid and Hormone Homeostasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Janne Hukkanen, Oulu University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Rifampisiini01
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: Glucose Tolerance
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifampicin (Active Comparator)
  Interventions: Drug: Rifampicin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifampicin
  Other Names: Rimapen, ATC J04AB02
  Arms: Rifampicin
Drug: Placebo
  Arms: Placebo

SUMMARY:
This clinical trial is designed to study the effects of rifampicin on the glucose, lipid and hormone homeostasis in healthy volunteers. The main hypothesis is that rifampicin lowers fasting glucose and enhances insulin sensitivity. The study is a randomized, placebo-controlled, open-label cross-over trial. Twelve subjects will be given 600 mg of rifampicin a day for a week compared to a one-week placebo arm. There is at least a 4-week wash-out between the arms. The main outcome measures are the changes in the fasting glucose and HOMA-IR-index (calculated based on fasting glucose and insulin).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Age 18-40 years

Exclusion Criteria:

* Any continuous medication
* Any significant disease
* Allergy to rifampicin
* Pregnancy and breast feeding
* Fear of needles and previous difficult blood samplings
* Substance abuse
* Participation in another clinical drug trial within 1 month of enrollment
* Use of soft contact lenses

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Fasting glucose

CONTACTS AND LOCATIONS:
Overall Officials: Janne Hukkanen, MD, PhD, Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Rahunen R, Kummu O, Koivukangas V, Hautajarvi H, Hakkola J, Rysa J, Hukkanen J. Pregnane X Receptor-4beta-Hydroxycholesterol Axis in the Regulation of Overweight- and Obesity-Induced Hypertension. J Am Heart Assoc. 2022 Mar 15;11(6):e023492. doi: 10.1161/JAHA.121.023492. Epub 2022 Mar 1. PMID 35229613